CLINICAL TRIAL: NCT00839124
Title: A Study of Inhalation of 20,000 EU Clinical Center Reference Endotoxin in Normal Volunteers Compared to Allergic Asthmatic Individuals
Brief Title: A Study of Inhalation of 20,000 EU CCRE in Normal Volunteers Compared to Allergic Asthmatic Individuals
Acronym: Endomac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08-1750 (CTRC # 2776); 5U19AI077437-02 (NIH)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Asthma; Hypersensitivity
Keywords: normal volunteer; healthy control volunteer; healthy subjects; asthma; allergy; allergic asthma
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Air Pollution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allergic asthma (Active Comparator): subjects with allergic asthma will undergo challenge with 20,000 EU CCRE
  Interventions: Biological: Clinical Center Reference Endotoxin (CCRE)
- healthy control (Active Comparator): Healthy volunteers will undergo challenge with 20,000 EU CCRE
  Interventions: Biological: Clinical Center Reference Endotoxin (CCRE)

INTERVENTIONS:
Biological: Clinical Center Reference Endotoxin (CCRE) — inhalation challenge with 20,000 EU CCRE
  Other Names: air pollution
  Arms: healthy control
Biological: Clinical Center Reference Endotoxin (CCRE) — inhalation of 20,000 EU CCRE
  Other Names: air pollution
  Arms: Allergic asthma

SUMMARY:
This will be a single center, open label study comparing baseline characteristics of recovered sputum cells (collected on screening day) to those of cells recovered 6 hours after inhalational challenge with 20,000 EU Clinical Center Reference Endotoxin (CCRE, a component of air pollution)) within each group as well as cross group comparisons between individuals with allergic asthma (AA's)and normal volunteers (NV's). The primary objective of this study is to test the hypothesis that persons with allergic asthma will have an increased neutrophil response to challenge with 20,000 EU CCRE compared to normal volunteers. Secondary objectives include post CCRE comparison between AA's and NV's with regard to changes in airway cells and blood as well as changes in mucociliary clearance (MCC) in response to inhalation of 20,000 EU CCRE.

DETAILED DESCRIPTION:
This will be a single center, open label study of allergic asthmatic and normal volunteers. The protocol will compare baseline characteristics of recovered sputum cells (collected on screening day) to those of cells recovered 6 hours after inhalational challenge with CCRE within each group as well as cross group comparisons between AA's and NV's. The following information indicates procedures to be performed at each visit as well as the anticipated duration of visits. Subsequent to this description are details regarding specific study procedures.

Visit 1: Baseline Visit (5 hours)

1. Consent will be obtained, review of subject's medical history, current medications and inclusion/exclusion criteria.
2. Vital sign measurements (temperature, pulse, respiratory rate, blood pressure), oxygen saturation, and symptom scoring
3. Urine pregnancy test for women of child bearing potential
4. Spirometry
5. Venipuncture for CBC with differential and baseline blood analyses
6. Physical exam of the ears, nose, throat and chest
7. Collection of exhaled breath for measurement of nitric oxide level
8. Xenon equilibrium gas scan and MCC
9. MCC scan
10. Sputum induction
11. After completion of the sputum induction, subjects will have brief MCC scan (< 10 minutes)

Visit 2: 24 hours post baseline subjects will return for the following 1 hour visit:

1. Review any change in medical status over prior 24 hours, vital signs, O2 saturation and symptom score
2. Follow up MCC scan

Visit 3: 24-48 hours prior to challenge visit at least 2 days after the baseline visit (½ hour)

1. Review change in medical status since last visit; vital signs, oxygen saturation, & symptom score
2. Urine pregnancy test
3. Spirometry

Visit 4: Endotoxin (CCRE) challenge day (8.5 to 9 hours)

1. Review any change in medical status since last visit
2. Vital signs, oxygen saturation, and symptom score
3. Spirometry
4. Physical exam of the ears, nose, throat and chest
5. If above measures are acceptable, CCRE challenge will be performed
6. Post-challenge monitoring including spirometry, vital signs, oxygen saturation, and symptom score at the following intervals post challenge: 30 and 60 minutes and then hourly for 5 additional hours.
7. Post challenge venipuncture (blood draw) for CBC with differential and post CCRE blood analyses
8. Collection of exhaled breath for measurement of nitric oxide level.
9. Four hours post challenge, subject will have MCC evaluated
10. After MCC is assessed, sputum induction will be performed.
11. After completion of the sputum induction, subjects will have brief MCC scan (< 10 minutes)
12. Discharge home or, alternatively, to GCRC for overnight observation per study MD.

Visit 5: 24 hours post challenge visit (1 hour)

1. Subject returns to the CEMALB, vital signs, oxygen saturation, and symptom score
2. Collection of exhaled breath for measurement of nitric oxide level.
3. Spirometry
4. Follow-up MCC scan
5. Each volunteer will be given a symptom scoring sheet for each day up to 96 hours (4 days) after challenge (see accompanying symptom scoring sheet in Appendix 3).

Post Challenge Observations/Reporting (5 minutes)

1. Subjects will be contacted for phone call follow-up 48-96 hours after challenge (see script Appendix 4 of accompanying protocol)

Study discontinuation visit within 10 days of the challenge dose: (15 minutes)

1. Vital signs, O2 saturation, symptom score, spirometry
2. If any findings are abnormal, medical evaluation as directed by the study physician will be undertaken Appendix 1 of the accompanying protocol provides a summary table regarding procedures performed at each subject study visit

ELIGIBILITY:
Inclusion Criteria for healthy controls:

* Normal lung function, defined as (Knudson 1976/1984 predicted set):

FVC of > 80 % of that predicted for gender, ethnicity, age and height FEV1 of > 80 % of that predicted for gender, ethnicity, age and height FEV1/FVC ratio of > .75

* Oxygen saturation of > 94 % and normal blood pressure (Systolic between 150 - 90, Diastolic between 90-60 mm Hg)
* Symptom Score no greater than 6 (out of a possible 24) for total symptom score with a value no greater than 2 for any one score.
* Negative methacholine inhalation challenge as performed in the screening protocol. (Less than a 20% decrease in FEV1 at a maximum methacholine concentration of 10 mg/ml)

  --Negative pregnancy test for females
* Negative allergy skin test (AST)

Inclusion criteria for allergic asthmatics also include:

* History of episodic wheezing, chest tightness, or shortness of breath after age of 6 years consistent with asthma, or physician diagnosed asthma after age of 6 years.
* Positive methacholine test.
* FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .70 (without use of bronchodilating medications for 12 hours)
* Allergic sensitization to at least one of the following allergen preparations: (House Dust Mite f, House dust mite p, Cockroach, Tree mix, Grass Mix, Weed Mix, Mold Mix 1, Mold Mix 2, Rat, Mouse, Guinea Pig, Rabbit, Cat or Dog) confirmed by positive AST.
* Negative allergy skin test as performed in the screening protocol.

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, or chronic thyroid disease.
* Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
* Use of systemic steroid therapy within the preceding 12 months for an asthma exacerbation. All use of systemic steroids in the last year will be reviewed by a study physician.
* Use of inhaled steroids, cromolyn or leukotriene inhibitors (montelukast or zafirlukast) except for use of cromolyn exclusively prior to exercise.
* Use of daily theophylline within the past month.
* Use of tricyclics and MAO inhibitors
* Pregnancy or nursing a baby.
* Cigarette smoking > 1 pack per month.
* Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Exacerbation of asthma more than 2x/week which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
* Viral upper respiratory tract infection within 2 weeks of challenge.
* Any acute infection requiring antibiotics within 2 weeks of challenge
* Receipt of LAIV (Live Attenuated Influenza Vaccine), also know as FluMist®, within the prior 14 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to test the hypothesis that persons with allergic asthma will have an increased neutrophil response to challenge with 20,000 EU CCRE compared to normal volunteers | 6 hours post challenge

SECONDARY OUTCOMES:
Secondary objectives include post CCRE comparison between AA's and NV's with regard to changes in airway cells and blood as well as changes in mucociliary clearance (MCC) in response to inhalation of 20,000 EU CCRE. | 6-24 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Bennett WD, Alexis NE, Almond M, Herbst M, Zeman KL, Peden DB. Effect of inhaled endotoxin on mucociliary clearance and airway inflammation in mild smokers and nonsmokers. J Aerosol Med Pulm Drug Deliv. 2014 Dec;27(6):459-65. doi: 10.1089/jamp.2013.1089. PMID 24568613
- [Derived] Bennett WD, Herbst M, Zeman KL, Wu J, Hernandez ML, Peden DB. Effect of inhaled endotoxin on regional particle deposition in patients with mild asthma. J Allergy Clin Immunol. 2013 Mar;131(3):912-3. doi: 10.1016/j.jaci.2012.09.010. Epub 2012 Oct 25. No abstract available. PMID 23102735